CLINICAL TRIAL: NCT03088696
Title: Evaluation of PC 6 "Neiguan" With Conventional Acupuncture to Prevent PONV After Laparoscopic Cholecystectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Data Nurse, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Neiguan PC6
Record Dates: First submitted 2017-03-07; First posted 2017-03-23 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Cholecystitis; Vomiting; Nausea
Keywords: laparoscopic; acupuncture
MeSH Terms: conditions — Cholecystitis; Vomiting; Nausea

STUDY DESIGN:
Intervention Model Description: randomized comparative double blind prospective study
Who Masked: Participant, Outcomes Assessor
Masking Description: The care provider get's an envelope from the study nurse when going to the patient in the operating room. Only the study nurse knows if an acupuncture needle is in the envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- stimulation of the acupuncture point (Active Comparator): a acupuncture needle and bandage will be applied at pericardium channel 6, point "Neiguan"
  Interventions: Other: stimulation
- no stimulation of the acupuncture point (Placebo Comparator): only a bandage will be applied at pericardium channel 6, point "Neiguan"
  Interventions: Other: no stimulation

INTERVENTIONS:
Other: stimulation — activation of the acupuncture point
  Arms: stimulation of the acupuncture point
Other: no stimulation — no activation of the acupuncture point
  Arms: no stimulation of the acupuncture point

SUMMARY:
Assessment of the effectiveness of PC 6 "Neiguan" with conventional acupuncture for preventing PONV (PostOperative Nausea and Vomiting) after laparoscopic surgery.

DETAILED DESCRIPTION:
Utilizing acustimulation, the effect of PC 6 "Neiguan" (acupuncture point Pericardium 6) has been studied in PONV . Conventional acupuncture has not been tested yet in laparoscopic cholecystectomy.

The incidence of postoperative vomiting during the first 24 hours is the main outcome. Secondary outcomes include: complete response rate, total rescue ondansetron dose used and patient satisfaction with PONV management.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients
* > 18 y
* General anesthesia
* Undergoing laparoscopic surgery
* Patient with American Society of Anesthesiologists physical status I-II
* Written informed consent

Exclusion Criteria:

* Pregnant women and breastfeeding
* Patient with cardiac disease
* Surgery more than 2 h
* No bowel surgery
* Signs of skin infection at or near the purposed site of the acupuncture point
* Patient with American Society of Anesthesiologists physical status IIII-IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Vomiting and Nausea | 24 hours
  numeric from 0-4, 0= no vomiting, 1= nausea, 2= moderate, 3= multiple and 4= extensive

SECONDARY OUTCOMES:
Use of antiemetic | 24 hours
  dosage in mg
Use of analgesia | 24 hours
  dosage in mg

CONTACTS AND LOCATIONS:
Overall Officials: Jan Poelaert, PhD MD, Study Chair — Universitair Ziekenhuis Brussel; Güngör Badaş, Nurse, Principal Investigator — Universitair Ziekenhuis Brussel; Vincent Van Tittelboom, MD, Study Director — Universitair Ziekenhuis Brussel; Philippe Bral, MD, Study Director — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No